CLINICAL TRIAL: NCT00630487
Title: Prospective, Randomized, Double Blind Placebo-Controlled Trial On The Efficacy Of Growth Hormone Replacement Therapy In Adult Patients With Isolated Growth Hormone Deficiency (PRO ISO-GHD Study)
Brief Title: Efficacy of Somatropin in Adult Patients With Isolated Growth Hormone Deficiency
Acronym: IGHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6281282
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2011-01-27 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Verum (Active Comparator)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Placebo — Patients of Placebo Group will be treated with placebo sub-cutaneous in the same way as Somatropin during the double blind treatment phase. To maintain blind subject will be measured in the same way as the treatment group for IGF-I- Levels. Central lab will randomize placebo patients to dose change or maintenance of dose. This will ensure continued blinding of the study to patients and personnel.
  Arms: Placebo
Drug: Somatropin — Fixed doses for patients: MALE: < 45y 0,4 mg, > 45y 0,2mg FEMALE: < 45y 0,5mg, >45y 0,3mg. for the first 4 weeks half of the dose will be given. After that dose will be increased to the targeted maintenance dose according to IGF-I Levels +/- 2 SD of age adjusted reference range. In case of side effects dosage will remain on half-dose (during the first 4 weeks) or reduced to half dose (after the first 4 weeks). At week 52 patients have the opportunity to switch to open label study restarting with half the given fixed dose which will be adjusted to full dose after 4 weeks.
  Arms: Verum

SUMMARY:
The study will investigate the effect on growth hormone replacement in patients with isolated growth hormone deficiency on body composition, especially visceral fat mass.

DETAILED DESCRIPTION:
The study was terminated on 15-Dec-2008 due to poor recruitment. Although 9 Patients were enrolled, no patient was randomized nor treated with somatropin. No safety reasons contributed to the termination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age
* Isolated growth hormone deficiency

Exclusion Criteria:

* Isolated growth hormone deficiency by childhood onset
* Diabetes mellitus type 1 or 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Pfizer Investigational Site, Bad Aibling
  - Pfizer Investigational Site, München

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281282&StudyName=Efficacy%20Of%20Somatropin%20In%20Patients%20With%20Isolated%20Growth%20Hormone%20Therapy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation and Completion Dates: 26 May 2008 to 17 October 2008. The study was terminated prematurely.
Pre-assignment Details: Nine patients were enrolled, but no patients were randomized due to early termination of study.
Groups:
- Somatropin: Growth hormone (GH) replacement therapy in fixed dose regimen according to age and gender: males less than or equal to 45 years receive 0.4 milligrams (mg) and females receive 0.5mg. Males greater than 45 years receive 0.2 mg and females receive 0.3 mg.
Period: Overall Study
Arm/Group | Placebo | Somatropin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Somatropin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Change of Visceral Fat Mass Assessed by Magnetic Resonance Imaging Scanning (MRI)
Description: Fat measurements carried out with the subjects lying in a supine position in a MRI scanner. Measurements of regional body fat obtained between the level of the coccygeal bone and the 2nd or 3rd lumbar vertebra.
Time Frame: Baseline, 52 weeks
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Visceral Fat Mass in Subgroups
Description: Change in visceral fat mass in subgroups. Subgroup 1: isolated GHD due to surgery and/or irradiation of pituitary adenoma and suprasellar tumors. Subgroup 2: history of traumatic brain injury (TBI) or subarachnoid hemorrhage (SAH).
Time Frame: Baseline, 52 weeks, 78 weeks
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Anthropometric Parameters (Height)
Time Frame: Baseline, 52 weeks, 78 weeks
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Anthropometric Parameters (Weight)
Time Frame: Baseline, 52 weeks, 78 weeks
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Anthropometric Parameters (Waist Circumference)
Time Frame: Baseline, 52 weeks, 78 weeks
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Alertness (Testbatterie Zur Aufmerksamkeitsprüfung [TAP]) and Memory (Auditory Verbal Learning Test [AVLT])
Description: Alertness: software-based neuropsychological assessment for response time and errors. Memory: analysis of learning and retention using 5-trial presentation of 15-word list (A), single presentation of interference list (B), 2 postinterference recall trials - 1 immediate, 1 delayed - and recognition of the target words with distractors (C). Performance variables were immediate word span under overload conditions, final acquisition level, amount learned in 5 trials, interference, delayed recall, and recognition (implicit learning).
Time Frame: Baseline, Week 52, Week 78
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Blood pressure was measured seated, the subject's arm supported at the level of the heart, and recorded to the nearest mm Hg. The same arm (preferably the dominant arm) was used throughout the trial. The subject was seated for 5 minutes before the blood pressure was obtained. Use of an automated device could have been used for measuring blood pressure.
Time Frame: Baseline, Week 52, Week 78
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Heart Rate
Description: The use of an automated device for measuring pulse rate was acceptable, although, when done manually, pulse rate was measured in the brachial/radial artery for at least 30 seconds.
Time Frame: Baseline, Week 52, Week 78
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Executive Function and Memory in Subgroups
Description: Change in executive function and memory in subgroups. Subgroup 1: isolated Growth Hormone Deficiency (GHD)due to surgery and/or irradiation of pituitary adenoma and suprasellar tumors. Subgroup 2: history of traumatic brain injury (TBI) or subarachnoid hemorrhage (SAH). Median reaction time, the total number of errors, the number of omissions and the number of false positive reactions.
Time Frame: Baseline, Week 52, Week 78
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Safety Laboratory Assessments
Description: Prespecified safety laboratory assessments evaluated for change or no change from baseline. Possible responses were Yes/No.
Time Frame: Baseline, Week 52, Week 78
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment (HOMA)-Index
Description: HOMA index is calculated by 1 of 2 methods: HOMA-Index = fasting insulin measured in microunits per milliliter (µU/ml) times fasting glucose measured in milligrams per deciliter mg/dl) divided by 405 or HOMA-Index = fasting insulin (µU/ml) times fasting glucose measured in millimoles per liter (mmol/l) divided by 22.5.
Time Frame: Baseline, Week 52, Week 78
Population: Study terminated, no subjects were treated.
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Quality of Life Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA)
Description: Participant self administered questionnaire consisting of 25 items that evoke yes or no answers. A score of 1 is given to each item affirmed and these are summed to give the total score. The maximum score is 25, which represents a poor quality of life. The minimum score is 0, which represents a good quality of life.
Time Frame: Baseline, Week 52, Week 78
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF36)
Description: Participant self administered questionnaire that measures each of the following eight health concepts: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); Mental Health (MH) as well as a reported Health Transition item (HT). Scale range 0 to 100, higher scores indicate a better health-related quality of life.
Time Frame: Baseline, Week 52, Week 78
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D)
Description: Participant self-administered questionnaire EQ-5D, a 2 part generic health status instrument. The first part consists of 5 descriptors of current health state: mobility, self care, usual activities, pain/discomfort and anxiety/depression. Scores are assigned on a three-level scale (1= no problem, 2= some problem, 3= extreme problem). The second part was an overall rating of the participant's current health state using a 20 cm Visual Analogue Scale (EQ-VAS) with endpoints labelled 'best imaginable health state' and 'worst imaginable health state'.
Time Frame: Baseline, Week 52, Week 78
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Cardiovascular Risk Factors
Description: Change in values of laboratory tests indicative of possible cardiovascular risk factors: high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides, N-terminal pro brain natriuretic peptide)
Time Frame: Baseline, Week 52, Week 78
Arm/Group | Placebo | Somatropin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Somatropin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.